CLINICAL TRIAL: NCT00945880
Title: A Phase 1b, Open Label Study of the Safety, Tolerability Pharmacokinetics and Pharmacodynamics of 100 mg Clemizole Hydrochloride Administered Orally Twice a Day for 28 Days Immediately Prior to Initiation of Treatment With HCV Standard of Care Therapy in Treatment-Naïve Subjects Chronically Infected With HCV
Brief Title: Safety and Tolerability Study of Clemizole Hydrochloride to Treat Hepatitis C in Subjects Who Are Treatment-Naive
Acronym: CLEAN-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eiger BioPharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EIG-101
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Hepatitis C
Keywords: HCV; Hepatitis C; Hepatitis
MeSH Terms: conditions — Hepatitis C; Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental Group (Experimental): clemizole hydrochloride, 100mg, BID
  Interventions: Drug: clemizole hydrochloride

INTERVENTIONS:
Drug: clemizole hydrochloride — Two 50 mg capsules containing clemizole hydrochloride are to be administered orally twice a day for 28 days for a total daily dose of 200 mg. Followed immediately by standard of care treatment consisting of interferon and ribavirin

SUMMARY:
The purpose of this study is to test the hypothesis that clemizole hydrochloride is safe and well tolerated when administered to subjects who are infected with hepatitis C virus and have not yet received treatment. This study will also examine how the virus and body respond to clemizole hydrochloride.

DETAILED DESCRIPTION:
This study is a phase 1b, open label study of four weeks of treatment with 100 mg po BID of clemizole hydrochloride administered immediately prior to the initiation of treatment with HCV standard of care therapy consisting of pegylated interferon and ribavirin in treatment-naïve subjects chronically infected with HCV genotype 1 or genotype 2. The duration of the study for each subject will be approximately 11 weeks (up to three week screening period, four week treatment period and four week safety follow-up period). The duration of the entire study is anticipated to be approximately four months (first subject in to last subject out). Pharmacokinetic sampling will be done at Day 1 and Day 28 of dosing. PK sampling will be conducted only on subjects who have consented to participate in the PK portion of this study. Participation in PK sampling is optional for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 18 to 55 years of age who are diagnosed with HCV by PCR
* HCV treatment-naïve patients who have already committed to undergo standard of care therapy (SOC) for HCV (pegylated interferon and ribavirin), and who wish to participate in a study immediately prior to the initiation of SOC
* Chronic hepatitis C infection, genotype 1 or genotype 2, two documented tests (PCR or HCV Ab; if one of the tests is HCV Ab, then the second test must be PCR and the PCR test must be at least 6 months after the HCV Ab test) at least 6 months apart
* Liver biopsy within the last two (2) years (biopsy can be done at the Screening Visit)
* Positive viral load of <1,000,000 IU/mL as measured by quantitative PCR
* Electrocardiogram (ECG) shows no acute ischemia or clinically significant abnormality and a QT/QTc interval <450 milliseconds - using Bazett's correction: QTc =QT/RR0.5 (ICH Guidance E14 Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs)
* Females of childbearing potential (intact uterus and within 1 year since the last menstrual period) should be non-lactating and have a negative serum pregnancy test. In addition, these subjects should agree to use one of the following acceptable birth control methods throughout the study:

  1. abstinence
  2. surgical sterilization (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) six months minimum
  3. IUD in place for at least six months
  4. barrier methods (condom or diaphragm) with spermicide
  5. surgical sterilization of the partner (vasectomy for six months)
  6. hormonal contraceptives for at least three months prior to the first dose of study drug
* Willing and able to comply with study procedures and provide written informed consent

Exclusion Criteria:

* Participation in a clinical trial with or use of any investigational agent within 30 days of Study Visit 1
* Patients co-infected with HIV
* Patients with screening tests positive for HBsAg, or anti-HIV Ab
* Liver biopsy within the last 2 years that shows Stage III fibrosis or higher
* Clinical evidence or suspicion of cirrhosis
* Active jaundice defined by total bilirubin >2.0
* INR ≥ 1.5
* Eating disorder or alcohol abuse within the past 2 years, excessive alcohol intake (>20 g per day for females (1.5 standard alcohol drinks) or >30 g per day for males (2.0 standard alcohol drinks) (a standard drink contains 14 g of alcohol: 12 oz of beer, 5 oz of wine or 1.5 oz of spirits) (1.0 fluid oz (US) = 29.57 ml), or if in the opinion of the investigator, an alcohol use pattern that will interfere with the study conduct
* Drug abuse within the last six months with the exception of cannabinoids and their derivatives
* Patients with absolute neutrophil count (ANC) <1500 cells/mm3; platelet count <135,000 cells/mm3; hemoglobin <12 g/dL for women and <13 g/dL for men; abnormal TSH,T4, or T3or thyroid function not adequately controlled; or serum creatinine concentration ≥1.5 times upper limit of normal (ULN)
* History or clinical evidence of any of the following:

  1. variceal bleeding, ascites, hepatic encephalopathy, CTP score >6, decompensated liver disease or any other form of non-viral hepatitis
  2. immunologically mediated disease (e.g., rheumatoid arthritis, inflammatory bowel disease, severe psoriasis, systemic lupus erythematosus) requiring more than intermittent nonsteroidal anti-inflammatory medications for management or that requires frequent or prolonged use of corticosteroids (inhaled asthma medications are allowed)
  3. any malignancy within 3 years except for basal cell skin cancer
  4. significant or unstable cardiac disease (e.g., angina, congestive heart failure, uncontrolled hypertension, history of arrhythmia)
  5. chronic pulmonary disease (e.g., chronic obstructive pulmonary disease) associated with functional impairment
  6. severe or uncontrolled psychiatric disease, including severe depression, history of suicidal ideation, suicidal attempts or psychosis requiring medication and/or hospitalization
* Patients with a body mass index >30 kg/m2
* Concomitant drugs known to prolong the QT interval (see Appendix E)
* Concomitant use of immunosuppressive or immune modulating agents
* Patients with any serious or condition that, in the opinion of the investigator, would preclude evaluation of response or make it unlikely that the contemplated course of therapy and follow-up could be completed or increase the risk to the subject of participation in the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the pharmacodynamic (PD) activity of a 100 mg po BID dose of clemizole hydrochloride on HCV viral load | Day 1, 3, 7, 14, 28, 56

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics (PK) of a 100 mg po BID dose of clemizole hydrochloride in subjects chronically infected with HCV | Day 1 and Day 28
Evaluate the safety and tolerability of four weeks of treatment with a 100 mg po BID dose of clemizole hydrochloride through review of adverse events | Day 1, 2, 3, 7, 14, 28, 56

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Glenn, MD, PhD, Study Director — Eiger BioPharmaceuticals, Inc.

REFERENCES:
- [Background] Einav S, Gerber D, Bryson PD, Sklan EH, Elazar M, Maerkl SJ, Glenn JS, Quake SR. Discovery of a hepatitis C target and its pharmacological inhibitors by microfluidic affinity analysis. Nat Biotechnol. 2008 Sep;26(9):1019-27. doi: 10.1038/nbt.1490. PMID 18758449